CLINICAL TRIAL: NCT04838431
Title: Development of a Prediction Model for Large for Gestational Age Infants at First Trimester: a Preliminary Study
Brief Title: A First Trimester Prediction Model for Large for Gestational Age Infants: a Preliminary Study
Acronym: PreMoLGA
Status: Terminated | Type: Observational
Why Stopped: Reached the sample size
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Prof. Fabio Facchinetti, Director of the Obstetrics and Gynecolocy department, University of Modena and Reggio Emilia
Other Study IDs: AOU: 0001395/20
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Large for Gestational Age Baby; Macrosomia, Fetal
Keywords: Prediction model; LGA; Singleton; Birtweight
MeSH Terms: conditions — Fetal Macrosomia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For each subject, blood sample is collected in fasting conditions for biochemical analyses of PAPP-A, PlGF, Inibin A, Insulin, high density lipoproteins (HDL) and triglycerides (TG), measured through routine laboratory methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample and ultrasound at first trimester — The blood sample and the ultrasound are part of the routine care for the aneuploidy screening at first trimester. We deepened the biochemicals and biophysical markers for predicting the risk for large for gestational age infants

SUMMARY:
Large for gestational age infants (LGA) have increased risks of adverse short-term perinatal outcomes. This study aims to develop a multivariable prediction model for the risk of giving birth to a LGA baby, by using biochemical, biophysical, anamnestic, and clinical maternal characteristics available at first trimester.

This prospective study includes all singleton pregnancies attending the first trimester aneuploidy screening at the Obstetric Unit of the University Hospital of Modena, in Northern Italy.

DETAILED DESCRIPTION:
For each subject, blood sample is collected in fasting conditions, then centrifuged, and the serum stored at minus 80° C, for subsequent biochemical analyses. PAPP-A, PlGF and Inibin A is measured with the automated DELFIA EXPRESS system (Thermo Fisher Scientific, Perkin Elmer ®). Insulin, high density lipoproteins (HDL) and triglycerides are measured through routine laboratory methods.

The mean arterial pressure (MAP) is measured with validated automated devices (Dinamap, BLTV6XX). After the women are seated and allowed to rest for 3-5 min, normal (22 to 32 cm) adult cuffs are fitted to their both arms. This is repeated two times with 1 min break in between. The MAP is calculated with the formula MAP DBP + 1/3(SBP - DBP) 21, where DBP represents diastolic blood pressure and SBP, systolic blood pressure. We calculate the final MAP as the average of all four measurements. Uterine artery Doppler studies including pulsatility index are measured through trans-abdominal ultrasound (Voluson E8 or Voluson E10) examinations. As indicated in Fetal Medicine Foundation (FMF), when carrying out Doppler studies, color flow mapping is used to identify each uterine artery along the side of the cervix and uterus at the level of the cervical internal os. Pulsed wave Doppler imaging is used with the sampling gate set at 2 mm to cover the whole vessel, and care is taken to ensure that the angle of insonation is less than 30°. When three to five similar consecutive waveforms are obtained, PI is measured. The uterine artery mPI is calculated by adding the right and left pulsatility index together, divided by two. All ultrasound and Doppler studies are carried out by a physician who had received the appropriate certificate of competence in the 11-13+6 week scans and Doppler study from the FMF.

Data on pregnancy outcome are collected from the hospital maternity records or directly from women if delivered elsewhere.

Medical records are reviewed by research associates to obtain anonymized data on mothers (i.e maternal demographics, BMI, age…) and their newborns (birthweight, gender, Apgar score, admission to the neonatal intensive care unit (NICU) and length of stay, neonatal morbidities, and mortality), and are organized in a password protected database.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies attending the first trimester Down syndrome screening at the University Hospital of Modena, in the North of Italy (tertiary Hospital).

Exclusion Criteria:

* Twin pregnancies
* Pregnancies with major fetal abnormalities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Singleton pregnancies attending the first trimester Down syndrome screening at the University Hospital of Modena, in the North of Italy (tertiary Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
LGA | From 37-42 weeks
  Risk for delivering a LGA infant, by combining the birtweight, the infant gender and the gestational age at birth

CONTACTS AND LOCATIONS:
Overall Officials: Fabio R Facchinetti, MD, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- University Hospital of Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We plan to validate the predictive model

REFERENCES:
- [Derived] Monari F, Menichini D, Spano' Bascio L, Grandi G, Banchelli F, Neri I, D'Amico R, Facchinetti F. A first trimester prediction model for large for gestational age infants: a preliminary study. BMC Pregnancy Childbirth. 2021 Sep 24;21(1):654. doi: 10.1186/s12884-021-04127-3. PMID 34560843